CLINICAL TRIAL: NCT01740375
Title: A Randomized Phase III Trial on the Role of Esophagectomy in Complete Responders to Preoperative Chemoradiotherapy for Squamous Cell Carcinoma of Esophagus
Brief Title: Role of Esophagectomy in Complete Responders to CCRT
Acronym: ESOPRESSO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: slow recruitment
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sung-Bae Kim, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Esophageal cancer AMC02
Record Dates: First submitted 2012-11-27; First posted 2012-12-04 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Esophagectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm B: observation: (No Intervention): No additional treatment after concurrent chemoradiotherapy. However, esophagectomy will be considered as a salvage treatment for local recurrence during observation.
- Arm A: esophagectomy (Experimental): Esophagectomy will be performed preferentially within 8 weeks (maximum 12 weeks) after completion of concurrent chemoradiotherapy
  Interventions: Procedure: esophagectomy

INTERVENTIONS:
Procedure: esophagectomy — esophagectomy
  Arms: Arm A: esophagectomy

SUMMARY:
To investigate the role of esophagectomy in complete responders to preoperative chemoradiotherapy for squamous cell carcinoma of esophagus, patients will be randomized to either observation or esophagectomy after concurrent chemoradiotherapy.

DETAILED DESCRIPTION:
After completion of concurrent chemoradiotherapy, patients will be reassed and visited to multidisciplinary clinic, then, randomized to either observation or esophagectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven squamous cell carcinoma of the intrathoracic esophagus
2. Surgically resectable (cT3, cT4a and/or disease with lymph node metastasis by AJCC 7th ed) esophageal cancer, as determined by Endoscopic Ultra Sound (EUS), chest CT and PET-CT
3. No prior treatment for the esophageal cancer
4. Age: 20-70 years
5. ECOG performance status 0, 1 or 2
6. Adequate hematological, renal, hepatic, pulmonary and cardiac functions defined as 6.1 Granulocytes > 1,500/microliter, Platelets > 75,000/microliter 6.2 Creatinine < 1.5 mg/dL (or CCr> 50 mg/mL), 6.3 Total bilirubin < 1.5 mg/dL 6.4 ALT and AST < 2.5 × upper normal limit 6.5 FEV1 >=1.5 L/min 6.6 Ejection fraction >= 45%
7. Non-pregnant, non-lactating female patients. Sexually active patients of childbearing potential must implement effective contraceptive practices during the study when treated with chemotherapy
8. Written, voluntary informed consent

Exclusion Criteria:

1. Subtypes other than squamous cell carcinoma
2. cT1N0M0, cT2N0M0 esophageal cancer or in situ carcinoma
3. Invasion of recurrent laryngeal, phrenic or sympathetic nerve
4. Invasion of the tracheobronchial tree or presence of tracheoesophageal fistula
5. Invasion of major vessels (vena cava, azygos vein and aorta) by the tumor
6. Malignant pleural effusion (documented by cytospin or cytology)
7. Cervical esophageal cancer
8. Para-aortic lymph node metastasis
9. Past or current history of malignancy other than entry diagnosis except for non-melanomatous skin cancer, curatively treated carcinoma in situ of the cervix, curatively treated early gastric cancer with endoscopic mucosal resection or a cured malignancy more than 5 years prior to enrollment
10. Previous chemotherapy or prior history of radiotherapy interfering with the planned radiotherapy as per protocol
11. Patients with a known history of HIV seropositivity or HCV (+). Patients with HBV (+) are eligible. However, primary prophylaxis using antiviral agents (i.e. lamivudine, etc) is recommended for HBV carrier to prevent HBV reactivation during whole treatment period.
12. Other serious illness or medical conditions A. Unstable cardiac disease (i.e. congestive heart failure, arrhythmia, symptomatic coronary artery disease) despite treatment, myocardial infarction within 6 months prior to study entry B. History of significant neurologic or psychiatric disorders including dementia or seizures C. Active uncontrolled infection (viral, bacterial or fungal infection) D. Other serious medical illnesses
13. New York heart Association Class III/IV and history of active angina. Documented myocardial infarction within the 6 months preceding registration. Patients with a history of significant ventricular arrhythmia requiring medication or congestive heart failure. History of 2nd or 3rd degree heart blocks.
14. Active infection or other serious underlying medical condition which would impair the ability of the patient to receive the planned treatment
15. Dementia or altered mental status that would prohibit the understanding and giving of informed consent
16. Uncontrolled diabetes mellitus: fasting glucose >150 mg/dL or patients requiring insulin therapy for glycemic control; fasting glucose >150 mg/dL or patients requiring insulin therapy for glycemic control;

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 486 (Estimated)
Dates: Start 2012-11; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
2-year disease-free survival (DFS) rate | 2 years from the enrollment of last patient

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years from the enrollment of last patient
progression-free survival | 5 years from the enrollment of last patient
failure pattern | 5 years from the enrollment of last patient
Number of Participants with Adverse Events | up to 60 days after treatment
Comparison of clinical complete response (cCR) vs. pathologic complete response rate (pCR) in patients who underwent esophagectomy | 5 years
Comparison of OS according to clinical response (CR vs PR vs SD/PD) after preoperative chemoradiotherapy among those who underwent preplanned esophagectomy; | 5 years from the enrollment of the last patient
Comparison of OS according to metabolic response after induction chemotherapy | 5 years from the enrollment of the last patient
Quality of life | 5 years from the enrollment of the last patient
Comparison of PFS according to clinical response (CR vs PR vs SD/PD) after preoperative chemoradiotherapy among those who underwent preplanned esophagectomy; | 5 years from the enrollment of the last patient
Comparison of TTF according to clinical response (CR vs PR vs SD/PD) after preoperative chemoradiotherapy among those who underwent preplanned esophagectomy; | 5 years from the enrollment of the last patient
Comparison of PFS according to metabolic response after induction chemotherapy | 5 years from the enrollment of the last patient
Comparison of TTF according to metabolic response after induction chemotherapy | 5 years from the enrollment of the last patient
treatment-related mortality | up to 60 days after completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Bae Kim, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Al-Batran SE, Koch C. Neoadjuvant therapy for oesophageal cancer: refining the armamentarium. Lancet. 2024 Jul 6;404(10447):5-7. doi: 10.1016/S0140-6736(24)01084-5. Epub 2024 Jun 11. No abstract available. PMID 38876135